CLINICAL TRIAL: NCT03842566
Title: Evaluation of Age-Related Skin Changes Using Clinical Probe Measurements and Imaging
Brief Title: Evaluation of Age-Related Skin Changes
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-602-000
Record Dates: First submitted 2019-01-24; First posted 2019-02-15 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Age-related Skin Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 20-29 Years Old
- 30-39 Years Old
- 40-49 Years Old
- 50-59 Years Old
- 60-69 Years Old
- 70-79 Years Old

SUMMARY:
This trial is a knowledge study utilizing skin measurement probes that are non-invasive instruments, with negligible risks for the subjects. No product will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects with Fitzpatrick skin type II or III.
* Subject agreeing to complete all study required procedures.
* Subject having given freely and expressly her informed consent.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or being in an exclusion period for a previous study.
* Subject who underwent tissue augmentation with dermal fillers including HA, calcium hydroxylapatite, autologous fat, mesotherapy, or other cosmetic procedures (eg, face-lift, laser, photomodulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, liposuction of the thigh, or other ablative procedures) in the face or thigh within 12 months before study entry or was planning to undergo any such treatment during the study.
* Subject who underwent treatment with botulinum toxins in the face or neck within 6 months of study entry or was planning to undergo such treatment during the study.
* Subject who ever received semi-permanent fillers or permanent facial implants (eg, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene) anywhere in the face or thigh, or was planning to be implanted with any of these products at any time during the study.
* Subject with current cutaneous inflammatory or infectious processes (eg, acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion on the face or thigh that could interfere with measurements.
* Subject having changed, started or stopped any hormonal treatment or any treatment likely to have an impact on skin condition (over-the-counter or prescription, oral or topical, or anti-wrinkle products on the face), within 30 days prior to enrollment or is planning to begin using such products during the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 100 female subjects will be included, with at least 10 subjects per age decade
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Age-related changes in fine lines on the cheek | 4 Months
  Measured using a 5 point photonumeric scale (Allergan Fine Lines scale)
  The scale range is 0 to 4, with 0 indicating no fine lines and 4 being the most severe fine lines (greater than 5 superficial lines with crosshatching).
Age-related changes in skin hydration on the cheek | 4 Months
  Tissue dielectric constant measurement using MoistureMeter D (Delfin Technologies). Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
Age-related changes in skin hydration on the cheek | 4 Months
  Tissue dielectric constant measurement using a Corneometer (Courage & Khazaka). Tissue dielectric constant is expressed as a unitless value that is directly proportional to the amount of water in the tissue.
Age-related changes in skin barrier function on the cheek | 4 Months
  Transepidermal water loss measurement using an AquaFlux AF100 (Biox Systems Ltd)
Age-related changes in skin radiance on the cheek | 4 Months
  Measurement of light reflection using a Skin-Glossymeter GL200 (Courage & Khazaka)
Age-related changes in skin color on the cheek | 4 Months
  Skin colorimetric measurement using a Spectrophotometer (Konica Minolta)
Age-related changes in skin melanin on the cheek | 4 Months
  Colorimetric measurement of skin melanin using a Mexameter MX18 (Courage & Khazaka)
Age-related changes in skin elasticity on the cheek and thigh | 4 Months
  Skin elasticity measurement using a Cutometer (Courage & Khazaka), ElastiMeter (Delfin Technologies), and Dermal Torque Meter (Dia-Stron Limited)
Age-related changes in skin thickness on the cheek and thigh | 4 Months
  Ultrasound imaging using a Dermascan Ultrasound (Cortex Technology)
Age-related changes in skin topography on the cheek and thigh | 4 Months
  Skin topography imaged using a PRIMOS (Canfield Scientific) fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rz (average height of roughness), and Rt (maximum height of the roughness profile).
Age-related changes in skin topography on the cheek and thigh | 4 Months
  Skin topography imaged using a DermaTOP (EOTECH) fringe projection imaging system. Output measurements from the images will include Ra (average roughness), Rz (average height of roughness), and Rt (maximum height of the roughness profile).
Age-related changes in skin density on the cheek and thigh | 4 Months
  Ultrasound imaging using a Dermascan Ultrasound (Cortex Technology)

SECONDARY OUTCOMES:
Reproducibility and repeatability of the skin hydration measurement on the cheek | 4 Months
  The reproducibility and repeatability of the tissue dielectric constant measurement using MoistureMeter D (Delfin Technologies) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the skin hydration measurement on the cheek | 4 Months
  The reproducibility and repeatability of the tissue dielectric constant measurement using a Corneometer (Courage & Khazaka) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the skin barrier function measurement on the cheek | 4 Months
  The reproducibility and repeatability of the Transepidermal water loss measurement using an AquaFlux AF100 (Biox Systems Ltd) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the skin radiance measurement on the cheek | 4 Months
  The reproducibility and repeatability of the light reflection using a Skin-Glossymeter GL200 (Courage & Khazaka) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the skin color measurement on the cheek | 4 Months
  The reproducibility and repeatability of the skin colorimetric measurement using a Spectrophotometer (Konica Minolta) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the skin melanin changes on the cheek | 4 Months
  The reproducibility and repeatability of the colorimetric measurement of skin melanin using a Mexameter MX18 (Courage & Khazaka) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the changes in skin elasticity on the cheek and thigh | 4 Months
  The reproducibility and repeatability of the skin elasticity measurement using a Cutometer (Courage & Khazaka), ElastiMeter (Delfin Technologies), and Dermal Torque Meter (Dia-Stron Limited) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the changes in skin thickness and density on the cheek and thigh | 4 Months
  The reproducibility and repeatability of the measurement of ultrasound imaging using a Dermascan Ultrasound (Cortex Technology) will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the changes in skin topography on the cheek | 4 Months
  The reproducibility and repeatability of the skin topographyusing a PRIMOS (Canfield Scientific) fringe projection imaging system will be determined by repeating the measurement three times by two technicians
Reproducibility and repeatability of the changes in skin topography on the cheek | 4 Months
  The reproducibility and repeatability of the skin topography will be imaged using a DermaTOP (EOTECH) fringe projection imaging system and will be determined by repeating the measurement three times by two technicians

CONTACTS AND LOCATIONS:
Overall Officials: Siham Rharbaoui, MD, Principal Investigator — DERMSCAN - Pharmascan
Locations (1):
- Dermscan-Pharmascan, Villeurbanne, France